CLINICAL TRIAL: NCT02914314
Title: An Open-Label Study With an Extension Phase to Evaluate the Pharmacokinetics of Perampanel (E2007) Oral Suspension When Given as an Adjunctive Therapy in Subjects From 1 Month to Less Than 4 Years of Age With Epilepsy
Brief Title: Pharmacokinetic Study With an Oral Suspension of Perampanel as Adjunctive Therapy in Pediatric Subjects With Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-G000-238
Record Dates: First submitted 2016-05-26; First posted 2016-09-26 (Estimated); Results first posted 2023-09-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-05

CONDITIONS: Epilepsy
Keywords: epilepsy; refractory partial seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Perampanel up to 12 or 16 mg/day (Experimental): Pediatric participants, ranging from 1 month to less than 4 years of age, will receive perampanel oral suspension once a day in titration period starting at Week 0 at a dose of 0.50 mg per day (mg/day) titrated up to 4 mg/day (for participants taking non-EIAED) or up to 8 mg/day (for participants taking EIAED). Depending on participants clinical response, tolerability and investigator's decision, dose can be up titrated to 6 mg/day (for participants taking non-EIAED) and up titrated to 8 mg/day (for participants taking EIAED). Dose titration must not exceed 12 mg/day (non-EIAED) and 16 mg/day (EIAED). Participants will continue taking the perampanel oral suspension at dose level achieved at end of titration period through maintenance period of core study and maintenance period of extension phase (Up to Week 52).
  Interventions: Drug: perampanel

INTERVENTIONS:
Drug: perampanel — oral suspension.
  Other Names: E2007

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of perampanel during the Maintenance Period of the Core Study following oral suspension administration given as an adjunctive therapy in pediatric participants from 1 month to less than 4 years of age with epilepsy.

DETAILED DESCRIPTION:
This is a multicenter, open-label study comprised of pretreatment, treatment (core study), and extension phases that is designed to evaluate the PK of an oral suspension of perampanel (maximum dose must not exceed 12 milligrams per day [mg /day] for participants taking non-enzyme-inducing antiepileptic drug [non-EIAED] or 16 mg/day for participants taking EIAED) when given as an adjunctive therapy in participants ranging from 1 month to less than 4 years of age with epilepsy. The Pretreatment Phase will last up to 2 weeks, during which participants will be assessed for their eligibility to participate in the study. The Treatment Phase will consist of 3 periods: Titration (12 [for participants taking non-EIAED] to 16 weeks [for participants taking EIAED]), Maintenance (4 weeks), and Follow-Up (4 weeks; only for those participants who complete the Maintenance Period but do not continue into the Extension Phase and those participants who discontinue study participation). Extension Phase: The Extension Phase will consist of 2 periods: Maintenance (32 weeks [for participants taking EIAED]; 36 weeks [for participants taking non-EIAED]) and Follow-Up (4 weeks).

The maximum total duration of treatment for each participant will be 52 weeks and the maximum total duration of the study for each participant will be 58 weeks (2 weeks Pretreatment+52 weeks of treatment+4 weeks Follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, from 1 month to less than 4 years of age (and of at least 36 weeks gestational age) at the time of consent
* Have a minimum weight of 4 kilograms (kg) (8.8 pounds [lb])
* Have a diagnosis of epilepsy with any type of seizure according to the International League Against Epilepsy's (ILAE) Classification of Epileptic Seizures (1981). Diagnosis should have been established at least 2 weeks (≤6 months of age) or 4 weeks (>6 months of age) before Visit 1, by clinical history and an electroencephalogram (EEG) that is consistent with epilepsy; normal interictal EEGs will be allowed provided that the participant meets the other diagnosis criterion (i.e., clinical history)
* Have had brain imaging (computed tomography [CT] or magnetic resonance imaging [MRI]) before Visit 1 that ruled out a progressive cause of epilepsy
* Have had 1 or more seizure(s) before Visit 1
* Currently being treated with a stable dose (i.e., unchanged for at least 5 half-lives) of 1 to a maximum of 4 antiepileptic drugs (AEDs) (at least 6, but not more than 8, in the age group of 1 to less than 24 months, and up to 13 subjects in the age group of 2 to less than 4 years, will be taking 1 EIAEDs [that is, carbamazepine (CBZ), oxcarbazepine (OXC), phenytoin (PHT), or eslicarbazepine (ESL)] out of the maximum of 4 AEDs. The remaining participants cannot be taking any EIAEDs).
* Have been on their current concomitant AED(s) with a stable dose for at least 2 weeks or 5 half-lives, whichever is longer, before Visit 1
* Must have discontinued all restricted medications (example, medications known to be inducers of cytochrome P450 3A) at least 2 weeks or 5 half-lives (whichever is longer) before Visit 1
* If entering the Extension Phase, must have completed the last visit of the Maintenance Period of the Core Study

Exclusion Criteria:

* Have a history of status epilepticus that required hospitalization during the 3 months before Visit 1
* Have seizures due to treatable medical conditions, such as those arising due to metabolic disturbances, toxic exposure, or an active infection
* Have epilepsy secondary to progressive central nervous system (CNS) disease or any other progressive neurodegenerative disease, including tumors
* Have had epilepsy surgery within 1 year of Visit 1
* Are scheduled and/or confirmed to have epilepsy surgery within 6 months after Visit 1
* Used intermittent rescue benzodiazepines (i.e., 1 to 2 doses over a 24-hour period considered one-time rescue) 2 or more times in the 2 weeks before Visit 1
* Current use of felbamate, or any evidence of ongoing hepatic or bone marrow dysfunction associated with prior felbamate treatment. (Prior use of felbamate must be discontinued at least 8 weeks before Visit 1.)
* Current use of vigabatrin or any evidence of clinically significant vision abnormality associated with prior vigabatrin treatment. (Prior use of vigabatrin must be discontinued at least 2 weeks before Visit 1.)
* Are on ketogenic diet regimen that has not been stable for at least 4 weeks before Visit 1
* Concomitant use of other drugs known to influence the CNS, (other than AEDs for epilepsy), where the dose has not been stabilized for at least 5 half-lives or 2 weeks, whichever is longer, before Visit 1
* Have any concomitant illnesses/co-morbidities that could severely affect the participant's safety or study conduct
* Have evidence of clinically significant disease (e.g., cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the investigator(s) could affect the participant's safety or study conduct
* Have clinically significant laboratory abnormalities or any clinically acute or chronic disease
* Have evidence of significant active hepatic disease. Stable elevation of liver enzymes, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) due to concomitant medication(s), will be allowed if they are less than 3 times the upper limit of normal (ULN)
* Have clinical evidence of significant active hematological disease; white blood cell (WBC) count ≤2500/ microliter (μL) (2.50 x 10^9/Liter [L]) or an absolute neutrophil count ≤1000/μL (1.00 x 10^9/L)
* Have conditions that may interfere with their participation in the study and/or with the PK of study drug
* Have participated in a study involving administration of an investigational drug or device within 4 weeks before Visit 1, or within approximately 5 half-lives of the previous investigational compound, whichever is longer
* Have recently (within 30 days before Visit 1) been exposed to perampanel in a clinical study or by prescription, and/or previous discontinuation from perampanel treatment due to adverse events related to perampanel
* Have a clinically significant ECG abnormality, including prolonged corrected QT interval (QTc) defined as >450 milliseconds (msec)
* Have had multiple drug allergies or a severe drug reaction to an AED(s), including dermatological (e.g., Stevens-Johnson syndrome), hematological, or organ toxicity reactions

Ages: 1 Month to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2023-04-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (17):
  - Children's Hospital Los Angeles, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - NW FL Clinical Research Group, LL-ClinEdge- PPDS, Gulf Breeze, Florida
  - Axcess Medical Research, Loxahatchee Groves, Florida
  - Pediatric Neurology PA, Orlando, Florida
  - Pediatric Epilepsy And Neurology Specialists, Tampa, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Carle Foundation Hospital, Urbana, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Children's Mercy Hospital, Kansas City, Missouri
  - Children's Hospital at Saint Peter's University Hospital, New Brunswick, New Jersey
  - Duke University Medical Center, Children's Health Center, Durham, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center PPDS, Winston-Salem, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Child Neurology Consultants of Austin, Austin, Texas
  - Road Runner Research, Ltd, San Antonio, Texas
- Children's Clinical University Hospital, Riga, Latvia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in the United States and Latvia from 20 February 2017 to 25 April 2023.
Pre-assignment Details: A total of 26 participants were screened and enrolled, of which 5 were screen failure and 21 participants received the study treatment.
Groups:
- Cohort 1, Age >=1 to <=6 Months: Perampanel: Participants of age range from greater than or equal to (>=) 1 month to less than or equal to (<=) 6 months received perampanel 0.5 milligrams (mg), oral suspension, before bedtime during Week 0 and then dose up titrated to a maximum of 12 milligram per day (mg/day) (for participants who are not taking any EIAED]), or titrated up to a maximum of 16 mg/day (for participants who are taking any EIAED). Dose titration was up to Week 12 for Non-EIAED participants and up to Week 16 for EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose up to 12 mg/day (for non-EIAED participants) or 16 mg/day (for EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase. All participants who completed Core Phase, entered Extension Phase, and continued their optimal perampanel dose in extension phase for up to Week 52. The total treatment duration of Core Phase was up to 16 weeks for non-EIAED participants or up to 20 weeks for EIAED participants, and total treatment duration of Extension Phase was up to 36 weeks for non-EIAED participants and 32 weeks for EIAED participants.
- Cohort 2, Age >6 to <=12 Months: Perampanel: Participants of age range from greater than (>) 6 to <=12 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to a maximum of 12 mg/day (for participants who are not taking any EIAED), or titrated up to a maximum of 16 mg/day (for participants who are taking any EIAED). Dose titration was up to Week 12 for Non-EIAED participants and up to Week 16 for EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose up to 12 mg/day (for non-EIAED participants) or 16 mg/day (for EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase. All participants who completed Core Phase, entered Extension Phase, and continued their optimal perampanel dose in extension phase for up to Week 52. The total treatment duration of Core Phase was up to 16 weeks for non-EIAED participants or up to 20 weeks for EIAED participants, and total treatment duration of Extension Phase was up to 36 weeks for non-EIAED participants and 32 weeks for EIAED participants.
- Cohort 3, Age >12 to <24 Months: Perampanel: Participants of age range from >12 to less than (<) 24 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to a maximum of 12 mg/day (for participants who are not taking any EIAED), or titrated up to a maximum of 16 mg/day (for participants who are taking any EIAED). Dose titration was up to Week 12 for Non-EIAED participants and up to Week 16 for EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose up to 12 mg/day (for non-EIAED participants) or 16 mg/day (for EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase. All participants who completed Core Phase, entered Extension Phase, and continued their optimal perampanel dose in extension phase for up to Week 52. The total treatment duration of Core Phase was up to 16 weeks for non-EIAED participants or up to 20 weeks for EIAED participants, and total treatment duration of Extension Phase was up to 36 weeks for non-EIAED participants and 32 weeks for EIAED participants.
- Cohort 4, Age >=24 to <48 Months: Perampanel: Participants of age range from >=24 to <48 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to a maximum of 12 mg/day (for participants who are not taking any EIAED), or titrated up to a maximum of 16 mg/day (for participants who are taking any EIAED). Dose titration was up to Week 12 for Non-EIAED participants and up to Week 16 for EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose up to 12 mg/day (for non-EIAED participants) or 16 mg/day (for EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase. All participants who completed Core Phase, entered Extension Phase, and continued their optimal perampanel dose in extension phase for up to Week 52. The total treatment duration of Core Phase was up to 16 weeks for non-EIAED participants or up to 20 weeks for EIAED participants, and total treatment duration of Extension Phase was up to 36 weeks for non-EIAED participants and 32 weeks for EIAED participants.
Period: Core Phase (Up to 20 Weeks)
Arm/Group | Cohort 1, Age >=1 to <=6 Months: Perampanel | Cohort 2, Age >6 to <=12 Months: Perampanel | Cohort 3, Age >12 to <24 Months: Perampanel | Cohort 4, Age >=24 to <48 Months: Perampanel
Started | 4 | 5 | 9 | 3
Participants Who Did Not Take EIAED | 4 | 3 | 5 | 1
Participants Who Took EIAED | 0 | 2 | 4 | 2
Completed | 4 | 5 | 8 | 1
Not Completed | 0 | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Inadequate Therapeutic Effect | 0 | 0 | 1 | 0
Period: Extension Phase (Up to 36 Weeks)
Arm/Group | Cohort 1, Age >=1 to <=6 Months: Perampanel | Cohort 2, Age >6 to <=12 Months: Perampanel | Cohort 3, Age >12 to <24 Months: Perampanel | Cohort 4, Age >=24 to <48 Months: Perampanel
Started | 4 (All participants who completed core phase entered extension phase.) | 5 (All participants who completed core phase entered extension phase.) | 8 (All participants who completed core phase entered extension phase.) | 1 (All participants who completed core phase entered extension phase.)
Completed | 4 | 5 | 6 | 1
Not Completed | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Participant choice | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAS) was the group of participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment.
Groups:
- Cohort 1, Age >=1 to <=6 Months: Perampanel: Participants of age range from >=1 month to <=6 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to a maximum of 12 mg/day (for participants who are not taking any EIAED), or titrated up to a maximum of 16 mg/day (for participants who are taking any EIAED). Dose titration was up to Week 12 for Non-EIAED participants and up to Week 16 for EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose up to 12 mg/day (for non-EIAED participants) or 16 mg/day (for EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase. All participants who completed Core Phase, entered Extension Phase, and continued their optimal perampanel dose in extension phase for up to Week 52. The total treatment duration of Core Phase was up to 16 weeks for non-EIAED participants or up to 20 weeks for EIAED participants, and total treatment duration of Extension Phase was up to 36 weeks for non-EIAED participants and 32 weeks for EIAED participants.
- Cohort 2, Age >6 to <=12 Months: Perampanel: Participants of age range from >6 to <=12 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to a maximum of 12 mg/day (for participants who are not taking any EIAED), or titrated up to a maximum of 16 mg/day (for participants who are taking any EIAED). Dose titration was up to Week 12 for Non-EIAED participants and up to Week 16 for EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose up to 12 mg/day (for non-EIAED participants) or 16 mg/day (for EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase. All participants who completed Core Phase, entered Extension Phase, and continued their optimal perampanel dose in extension phase for up to Week 52. The total treatment duration of Core Phase was up to 16 weeks for non-EIAED participants or up to 20 weeks for EIAED participants, and total treatment duration of Extension Phase was up to 36 weeks for non-EIAED participants and 32 weeks for EIAED participants.
- Cohort 3, Age >12 to <24 Months: Perampanel: Participants of age range from >12 to <24 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to a maximum of 12 mg/day (for participants who are not taking any EIAED), or titrated up to a maximum of 16 mg/day (for participants who are taking any EIAED). Dose titration was up to Week 12 for Non-EIAED participants and up to Week 16 for EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose up to 12 mg/day (for non-EIAED participants) or 16 mg/day (for EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase. All participants who completed Core Phase, entered Extension Phase, and continued their optimal perampanel dose in extension phase for up to Week 52. The total treatment duration of Core Phase was up to 16 weeks for non-EIAED participants or up to 20 weeks for EIAED participants, and total treatment duration of Extension Phase was up to 36 weeks for non-EIAED participants and 32 weeks for EIAED participants.
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Age >=1 to <=6 Months: Perampanel | Cohort 2, Age >6 to <=12 Months: Perampanel | Cohort 3, Age >12 to <24 Months: Perampanel | Cohort 4, Age >=24 to <48 Months: Perampanel | Total
Number analyzed (Participants) | 4 | 5 | 9 | 3 | 21
Age, Continuous [Mean (Standard Deviation); unit: months] | 5.5 (0.58) | 10.2 (0.84) | 18.8 (3.73) | 31.3 (4.16) | 16.0 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 7 | 1 | 13
  Male | 2 | 2 | 2 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 1 | 4
  Not Hispanic or Latino | 3 | 5 | 7 | 2 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 2
  White | 3 | 5 | 7 | 2 | 17
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Core Phase and Extension Phase: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAE was an adverse event (AE) that emerged during treatment, having been absent at pretreatment (Baseline); or re-emerged during treatment, having been present at pretreatment (Baseline) but stopped before treatment; or worsened in severity during treatment relative to the pretreatment state, when AE was continuous. SAE was any untoward medical occurrence that at any dose: Resulted in death; was life-threatening (meaning participant was at an immediate risk of death from AE as it occurred; this did not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death); Required inpatient hospitalization or prolongation of existing hospitalization; Resulted in persistent or significant disability/incapacity; Was a congenital anomaly/birth defect (in child of a participant who was exposed to the study drug).
Time Frame: Core Phase: From the first dose of study drug up to 4 weeks of follow up after the last dose in Core Phase (up to Week 24); Extension Phase: From end of Core Phase treatment up to 4 weeks of follow up after the last dose in Extension Phase (up to Week 56)
Population: The SAS was the group of participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel: Participants of age range from >=1 month to <=6 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to a maximum of 12 mg/day (for participants who are not taking any EIAED), or titrated up to a maximum of 16 mg/day (for participants who are taking any EIAED). Dose titration was up to Week 12 for Non-EIAED participants and up to Week 16 for EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose up to 12 mg/day (for non-EIAED participants) or 16 mg/day (for EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase. The total treatment duration of Core Phase was up to 16 weeks for non-EIAED participants or up to 20 weeks for EIAED participants.
- Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel: Participants of age range from >6 to <=12 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to a maximum of 12 mg/day (for participants who are not taking any EIAED), or titrated up to a maximum of 16 mg/day (for participants who are taking any EIAED). Dose titration was up to Week 12 for Non-EIAED participants and up to Week 16 for EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose up to 12 mg/day (for non-EIAED participants) or 16 mg/day (for EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase. The total treatment duration of Core Phase was up to 16 weeks for non-EIAED participants or up to 20 weeks for EIAED participants.
- Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel: Participants of age range from >12 to <24 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to a maximum of 12 mg/day (for participants who are not taking any EIAED), or titrated up to a maximum of 16 mg/day (for participants who are taking any EIAED). Dose titration was up to Week 12 for Non-EIAED participants and up to Week 16 for EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose up to 12 mg/day (for non-EIAED participants) or 16 mg/day (for EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase. The total treatment duration of Core Phase was up to 16 weeks for non-EIAED participants or up to 20 weeks for EIAED participants.
- Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel: Participants of age range from >=24 to <48 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to a maximum of 12 mg/day (for participants who are not taking any EIAED), or titrated up to a maximum of 16 mg/day (for participants who are taking any EIAED). Dose titration was up to Week 12 for Non-EIAED participants and up to Week 16 for EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose up to 12 mg/day (for non-EIAED participants) or 16 mg/day (for EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase. The total treatment duration of Core Phase was up to 16 weeks for non-EIAED participants or up to 20 weeks for EIAED participants.
- Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel: Participants of age range from >=1 month to <=6 months who completed the Core Phase continued their optimal perampanel oral suspension, at the dose level achieved at the end of the Core Phase. The maximum total daily allowed dose for a non-EIAED participants was 12 mg and 16 mg for EIAED participants. The total treatment duration of Extension Phase was up to 36 weeks for non-EIAED participants and 32 weeks for EIAED participants.
- Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel: Participants of age range from >6 to <=12 months who completed the Core Phase continued their optimal perampanel oral suspension, at the dose level achieved at the end of the Core Phase. The maximum total daily allowed dose for a non-EIAED participants was 12 mg and 16 mg for EIAED participants. The total treatment duration of Extension Phase was up to 36 weeks for non-EIAED participants and 32 weeks for EIAED participants.
- Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel: Participants of age range from >12 to <24 months who completed the Core Phase continued their optimal perampanel oral suspension, at the dose level achieved at the end of the Core Phase. The maximum total daily allowed dose for a non-EIAED participants was 12 mg and 16 mg for EIAED participants. The total treatment duration of Extension Phase was up to 36 weeks for non-EIAED participants and 32 weeks for EIAED participants.
- Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel: Participants of age range from >=24 to <48 months who completed the Core Phase continued their optimal perampanel oral suspension, at the dose level achieved at the end of the Core Phase. The maximum total daily allowed dose for a non-EIAED participants was 12 mg and 16 mg for EIAED participants. The total treatment duration of Extension Phase was up to 36 weeks for non-EIAED participants and 32 weeks for EIAED participants.
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 4 | 5 | 9 | 3 | 4 | 5 | 8 | 1
Participants
  Participants with TEAEs | 3 | 5 | 9 | 3 | 4 | 5 | 8 | 1
  Participants with SAEs | 2 | 1 | 2 | 1 | 3 | 1 | 3 | 0

2. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Hematology Laboratory Parameters: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils, and Platelets
Description: Basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils, and platelets were expressed as 10^9 cells per liter (/L). Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameters was reported.
Time Frame: Core Phase: Baseline, end of Core Phase treatment (up to Week 20); Extension Phase: Baseline (Core Phase), end of Extension Phase treatment (Week 52)
Population: The SAS was the group of participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment. Here, "overall number of participants analyzed" signifies participants who were evaluable for this OM and "number analyzed" signifies participants who were evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 3 | 5 | 7 | 2 | 3 | 5 | 6 | 1
10^9 cells/L
  Change in Basophils | 0.03 (0.058) | -0.02 (0.110) | -0.06 (0.151) | 0.00 (0.000) | 0.03 (0.058) | 0.04 (0.219) | -0.05 (0.122) | 0.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Eosinophils | -0.03 (0.115) | -0.00 (0.100) | -0.04 (0.513) | -0.15 (0.212) | 0.10 (0.100) | 0.02 (0.148) | -0.05 (0.399) | 0.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Leukocytes | 1.73 (2.316) | 1.26 (5.855) | 1.10 (3.062) | 2.82 (6.187) | 2.43 (1.601) | -0.76 (4.558) | -1.08 (4.712) | -1.45 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Lymphocytes | 1.00 (1.500) | 0.62 (2.448) | 0.54 (2.099) | -1.73 (0.813) | 0.53 (0.757) | -0.24 (1.627) | -1.38 (2.555) | -1.75 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Monocytes | -0.13 (0.153) | 0.10 (0.308) | 0.10 (0.606) | 0.33 (0.672) | 0.10 (0.100) | -0.10 (0.292) | -0.02 (0.325) | 0.25 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Neutrophils | 0.90 (0.781) | 0.60 (3.820) | 0.51 (1.975) | 4.35 (6.435) | 1.70 (0.954) | -0.46 (2.518) | 0.38 (3.019) | 0.10 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Platelets: number analyzed (Participants) | 2 | 5 | 4 | 2 | 2 | 5 | 5 | 1
  Change in Platelets | -44.00 (108.894) | -63.80 (192.587) | 63.00 (167.127) | -22.50 (57.276) | 7.50 (98.288) | -32.00 (280.306) | 23.80 (147.041) | -85.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

3. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Hematology Laboratory Parameter: Erythrocytes
Description: Erythrocytes was expressed as 10^12 cells/L. Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameter was reported.
Time Frame: as for outcome 2
Population: The SAS was the group of participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment. Here, "overall number of participants analyzed" signifies participants who were evaluable for this OM.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 3 | 5 | 7 | 2 | 3 | 5 | 6 | 1
10^12 cells/L | 0.44 (0.576) | 0.16 (0.501) | 0.10 (0.155) | -0.10 (0.283) | 0.27 (0.329) | 0.39 (0.919) | -0.14 (0.396) | -0.03 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

4. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Hematology Laboratory Parameter: Hemoglobin
Description: Hemoglobin was expressed as grams per liter (g/L). Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameter was reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 3 | 5 | 7 | 2 | 3 | 5 | 6 | 1
g/L | 14.00 (18.000) | 5.20 (8.899) | 3.14 (3.237) | -0.25 (3.889) | 10.00 (8.888) | 12.80 (20.945) | -1.33 (13.808) | -6.50 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

5. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Clinical Chemistry Laboratory Parameters: Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Gamma Glutamyl Transferase, Lactate Dehydrogenase
Description: Alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, gamma glutamyl transferase, lactate dehydrogenase were expressed as units per liter (U/L). Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameters was reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 4 | 5 | 7 | 2 | 4 | 5 | 7 | 1
U/L
  Change in Alanine Aminotransferase | -2.25 (7.932) | -16.00 (27.803) | -13.71 (33.265) | 6.00 (15.556) | 36.50 (90.820) | -16.00 (27.313) | -11.43 (37.228) | -4.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Alkaline Phosphatase | 43.50 (115.610) | 266.00 (652.320) | 23.86 (21.162) | -46.50 (53.033) | -12.75 (97.072) | -32.40 (147.179) | -77.29 (205.368) | -58.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Aspartate Aminotransferase | -2.00 (2.449) | -12.20 (21.993) | -6.57 (16.009) | 0.50 (3.536) | 21.00 (58.980) | -13.20 (22.477) | -8.43 (19.569) | 1.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Gamma Glutamyl Transferase | 12.50 (87.577) | -3.00 (3.536) | -15.71 (31.653) | 5.00 (5.657) | 50.00 (320.278) | -5.40 (4.336) | -23.71 (48.801) | -1.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Lactate Dehydrogenase | -6.00 (50.721) | -32.60 (54.574) | -14.43 (28.425) | 51.50 (132.229) | 1.00 (68.775) | -44.60 (49.863) | -17.29 (67.037) | -39.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

6. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Clinical Chemistry Laboratory Parameter: Bilirubin
Description: Bilirubin was expressed as micromoles per liter (mcmol/L). Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameter was reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 4 | 5 | 7 | 2 | 4 | 5 | 7 | 1
mcmol/L | -0.30 (0.600) | 0.64 (2.057) | -0.46 (1.555) | 0.70 (0.990) | -0.10 (0.200) | 1.24 (2.414) | -0.57 (1.093) | 0.90 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

7. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Clinical Chemistry Laboratory Parameters: Calcium, Chloride, Cholesterol, Glucose, Phosphate, Potassium, Sodium, Triglycerides, Urea Nitrogen
Description: Calcium, chloride, cholesterol, glucose, phosphate, potassium, sodium, triglycerides, urea nitrogen were expressed as millimoles per liter (mmol/L). Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameters was reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 4 | 5 | 7 | 2 | 4 | 5 | 7 | 1
mmol/L
  Change in Calcium | -0.08 (0.147) | 0.02 (0.095) | -0.00 (0.098) | -0.01 (0.014) | -0.05 (0.123) | 0.05 (0.139) | -0.02 (0.103) | -0.04 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Chloride | -0.25 (2.500) | -0.80 (1.304) | -1.71 (3.450) | -1.00 (2.828) | 0.00 (2.160) | -2.60 (3.578) | 0.43 (1.988) | 1.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Cholesterol | 0.45 (0.191) | 0.52 (1.102) | -0.02 (0.505) | 0.58 (0.311) | -0.55 (0.583) | 1.48 (1.369) | 0.19 (0.578) | 0.83 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Glucose: number analyzed (Participants) | 2 | 4 | 2 | 0 | 2 | 4 | 5 | 0
  Change in Glucose | -0.42 (0.898) | 0.78 (0.668) | -0.24 (1.450) |  | 0.34 (1.096) | 0.18 (0.249) | -0.07 (0.640) |
  Change in Phosphate: number analyzed (Participants) | 4 | 2 | 7 | 2 | 4 | 2 | 7 | 1
  Change in Phosphate | -0.22 (0.277) | 0.11 (0.339) | -0.00 (0.154) | -0.31 (0.714) | 0.05 (0.169) | 0.16 (0.042) | -0.08 (0.145) | 0.07 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Potassium | -0.23 (0.222) | 0.06 (0.167) | 0.19 (0.652) | 0.25 (0.212) | -0.10 (0.712) | -0.02 (0.669) | 0.21 (0.285) | -0.60 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Sodium | 1.25 (2.986) | 0.00 (2.236) | -1.86 (2.911) | 4.00 (4.243) | 0.50 (3.109) | -0.40 (2.408) | 1.14 (0.690) | -2.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Triglycerides | 0.94 (0.619) | -0.50 (0.641) | 0.27 (1.047) | 0.44 (0.156) | 0.54 (0.602) | -0.05 (0.910) | -0.09 (0.544) | 0.05 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Urea Nitrogen | 0.27 (0.791) | 0.74 (1.440) | -0.97 (1.296) | 0.18 (1.768) | 1.69 (0.942) | 0.89 (3.316) | 0.61 (1.694) | 0.36 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

8. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Clinical Chemistry Laboratory Parameters: Creatinine, Direct Bilirubin, Urate
Description: Creatinine, direct bilirubin, urate were expressed as micromoles per liter (mcmol/L). Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameters was reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 4 | 5 | 7 | 2 | 4 | 5 | 7 | 1
mcmol/L
  Change in Creatinine | 2.25 (4.505) | 1.80 (4.024) | -1.28 (3.402) | 4.51 (6.357) | 6.51 (8.187) | 3.61 (4.929) | 1.29 (3.400) | 9.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Direct Bilirubin | 0.00 (0.000) | 0.08 (0.183) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.08 (0.183) | 0.00 (0.000) | 0.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Urate | 0.00 (0.024) | -0.02 (0.064) | -0.02 (0.032) | 0.01 (0.097) | -0.01 (0.054) | 0.01 (0.086) | -0.00 (0.045) | 0.04 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

9. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Clinical Chemistry Laboratory Parameters: Albumin, Globulin, Protein
Description: Albumin, globulin, protein were expressed as g/L. Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameters was reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 4 | 5 | 7 | 2 | 4 | 5 | 7 | 1
g/L
  Change in Albumin | 0.50 (1.291) | 2.00 (4.183) | -0.29 (2.059) | -1.00 (4.243) | 2.00 (3.266) | 5.60 (7.335) | -0.29 (2.870) | 2.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Globulin | 2.50 (6.455) | -2.20 (3.114) | 0.71 (1.496) | -2.00 (2.828) | 7.25 (8.057) | 0.20 (3.347) | 3.43 (2.760) | 3.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Protein | 3.00 (5.657) | -0.20 (2.588) | 0.43 (3.047) | -3.00 (7.071) | 9.25 (9.287) | 5.80 (7.596) | 3.14 (3.934) | 5.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

10. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Vital Sign Parameters: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured after the participant sitting or supine, for 5 minutes. SBP and DBP were expressed as millimeter of mercury (mmHg). Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameters was reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 3 | 5 | 9 | 3 | 3 | 5 | 8 | 1
mmHg
  Change in SBP | -1.00 (26.211) | 0.60 (6.066) | 0.33 (19.780) | 10.33 (4.726) | 27.00 (30.199) | 4.00 (5.477) | 10.63 (20.333) | 16.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in DBP | -5.33 (3.786) | 4.40 (5.857) | -0.89 (10.659) | 8.67 (6.429) | 23.00 (20.298) | 1.60 (5.941) | 6.00 (9.885) | 0.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

11. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Vital Sign Parameter: Pulse Rate
Description: Pulse rate measured after the participant sitting or supine, for 5 minutes and was expressed in beats per minute (beats/min). Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameter was reported.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 4 | 5 | 9 | 3 | 4 | 5 | 8 | 1
beats/min | 5.25 (16.112) | -4.40 (7.537) | -14.89 (14.675) | -21.67 (21.127) | -9.25 (14.773) | -15.80 (11.670) | -13.75 (9.543) | -26.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

12. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Vital Sign Parameter: Respiratory Rate
Description: Respiratory rate was the number of breaths taken per minute, measured at rest. Respiratory rate was expressed as breaths per minute (breaths/min). Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameter was reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 3 | 5 | 9 | 3 | 3 | 5 | 8 | 1
breaths/min | -5.33 (6.110) | -3.00 (4.183) | -4.78 (8.243) | -5.33 (2.309) | -4.33 (7.506) | -4.80 (5.541) | -3.88 (7.415) | 6.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

13. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Vital Sign Parameter: Body Temperature
Description: Body temperature was expressed as degree centigrade. Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameter was reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degree centigrade
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 3 | 5 | 9 | 3 | 3 | 5 | 8 | 1
degree centigrade | 0.10 (0.265) | -0.02 (0.130) | 0.02 (0.199) | 0.13 (0.153) | 0.47 (0.702) | 0.02 (0.045) | -0.16 (0.311) | -0.20 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

14. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Height
Description: Height was expressed as centimeters. Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameters was reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 4 | 5 | 9 | 2 | 4 | 5 | 8 | 1
centimeters | 4.76 (2.197) | 5.20 (2.361) | 5.06 (1.429) | 3.63 (1.237) | 17.65 (3.643) | 12.78 (2.548) | 10.24 (1.849) | 6.50 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

15. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Weight
Description: Weight was expressed as kilograms. Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameter was reported.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 4 | 5 | 9 | 3 | 4 | 5 | 8 | 1
kilograms | 1.88 (0.377) | 1.20 (1.065) | 1.01 (1.134) | 0.77 (0.153) | 3.88 (2.081) | 3.24 (1.356) | 2.88 (1.792) | 0.90 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

16. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Head Circumference
Description: Head circumference was expressed as centimeters. Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameter was reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 4 | 5 | 9 | 2 | 4 | 5 | 8 | 1
centimeters | 1.87 (1.231) | 1.50 (1.061) | 1.14 (1.927) | -0.15 (0.495) | 4.02 (0.846) | 2.50 (0.791) | 2.36 (1.537) | 0.50 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

17. Secondary Outcome: Core and Extension Phase: Mean Change From Baseline in ECG Parameters: Single Beat Heart Rate-corrected QT Interval (QTcB), QT Interval Corrected According to the Formula of Fridericia (QTcF), PR and QT Intervals, QRS Duration, and Aggregate RR Interval
Description: QTc: time from beginning of QRS complex to end of T wave, corrected for heart rate. QT interval: time from ECG Q wave to end of T wave corresponding to electrical systole. QRS interval: time from ECG Q wave to end of S wave, corresponding to ventricle depolarization. PR interval: time between beginning of P wave and start of QRS interval, corresponding to end of atrial depolarization and onset of ventricular depolarization. RR interval: time elapsed between two successive R waves of QRS signal. Single beat QTcB, QTcF, PR and QT Interval, QRS duration and aggregate RR interval were expressed as millisecond (msec). Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameters was reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 4 | 5 | 9 | 3 | 4 | 5 | 7 | 1
msec
  Change in Single Beat QTcB Interval: number analyzed (Participants) | 4 | 5 | 8 | 3 | 4 | 5 | 6 | 1
  Change in Single Beat QTcB Interval | -9.0 (24.06) | -7.0 (26.29) | -3.8 (33.86) | 17.0 (14.42) | -29.75 (27.476) | -5.60 (32.168) | 4.33 (8.710) | 58.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Single Beat QTcF Interval: number analyzed (Participants) | 4 | 5 | 8 | 3 | 4 | 5 | 6 | 1
  Change in Single Beat QTcF Interval | -4.5 (20.86) | -10.0 (21.99) | 1.9 (29.95) | 5.7 (8.62) | -8.25 (22.721) | -2.40 (36.115) | 1.17 (9.347) | 27.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Single Beat PR Interval: number analyzed (Participants) | 4 | 5 | 8 | 3 | 4 | 5 | 6 | 1
  Change in Single Beat PR Interval | -2.8 (4.57) | -2.8 (8.47) | -1.1 (16.66) | -10.3 (12.66) | 3.00 (3.162) | 3.80 (13.236) | 2.50 (8.689) | -3.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Single Beat QRS Duration: number analyzed (Participants) | 4 | 5 | 8 | 3 | 4 | 5 | 6 | 1
  Change in Single Beat QRS Duration | -0.5 (5.45) | -0.2 (5.89) | -0.8 (3.20) | -6.0 (8.00) | 3.75 (2.986) | -1.20 (6.181) | -1.67 (3.830) | 1.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Aggregate RR Interval | 28.3 (35.36) | -30.4 (26.37) | 60.7 (61.84) | -76.7 (77.36) | 165.25 (31.127) | 23.00 (72.087) | 20.57 (81.506) | -178.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Single Beat QT Interval: number analyzed (Participants) | 4 | 5 | 8 | 3 | 4 | 5 | 6 | 1
  Change in Single Beat QT Interval | 1.8 (17.23) | -13.8 (16.04) | 10.6 (29.61) | -10.0 (18.33) | 23.25 (14.569) | 2.40 (41.374) | -3.17 (15.779) | -16.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

18. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in ECG Parameter: ECG Ventricular Rate
Description: Ventricular rate is determined by dividing 60 by the mean RR interval of the ECG in seconds (mean time between QRS complexes) to get beats per minute. ECG ventricular rate was expressed as beats/min. Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameter was reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 4 | 5 | 9 | 3 | 4 | 5 | 7 | 1
beats/min | -7.5 (9.04) | 8.6 (7.37) | -12.2 (11.39) | 18.7 (22.85) | -36.25 (4.272) | -4.40 (15.437) | -3.14 (17.837) | 50.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

19. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Thyroid Stimulating Hormone (TSH): Thyrotropin
Description: Thyrotropin was expressed as milli-international units per liter (mIU/L). Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameter was reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 3 | 3 | 5 | 1 | 4 | 5 | 6 | 1
mIU/L | 1.12 (1.242) | -1.02 (0.279) | 1.33 (1.283) | -0.90 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis. | 0.05 (0.590) | -0.89 (1.405) | -0.08 (1.026) | -0.35 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

20. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Insulin-like Growth Factor 1 (IGF-1)
Description: IGF-1 was expressed as millimoles per liter*10^-6 (mmol/L*10^-6). Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameter was reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L*10^-6
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 1 | 3 | 5 | 1 | 3 | 4 | 7 | 1
mmol/L*10^-6 | -2.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis. | 7.00 (3.606) | 3.60 (6.066) | 1.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis. | 6.00 (0.000) | 4.75 (5.439) | 6.29 (9.160) | -1.00 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

21. Secondary Outcome: Core Phase and Extension Phase: Mean Change From Baseline in Free Thyroxine, and Free Triiodothyronine
Description: Free thyroxine, and free triiodothyronine were expressed as picomoles per liter (pmol/L). Change from baseline was calculated as post-baseline absolute value minus baseline value. Baseline values of Core Phase was used to calculate the change from baseline data for Extension Phase. Mean change from baseline data at end of Core Phase and at end of Extension Phase treatment for specified parameters was reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
Number analyzed (Participants) | 3 | 1 | 5 | 1 | 4 | 3 | 5 | 1
pmol/L
  Change in Free Thyroxine | 0.90 (1.931) | -1.30 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis. | -1.80 (1.147) | -3.90 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis. | 2.55 (1.021) | 0.83 (1.443) | 0.00 (0.919) | -3.90 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.
  Change in Free Triiodothyronine | -0.40 (0.889) | 0.60 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis. | 0.06 (0.885) | -4.30 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis. | 0.28 (1.250) | 1.03 (0.611) | -0.16 (1.230) | -1.80 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

22. Primary Outcome: Dose Normalized Area Under the Concentration-Time Curve for Dosing Interval at Steady State (AUCtau,ss) of Perampanel During the Maintenance Period of the Core Phase for Non-EIAED Participants
Description: Dose normalized AUCtau,ss was calculated as AUCtau,ss/maintenance dose, where AUCtau,ss is the area under the curve during a dosing interval (tau, 24 hours) at steady state calculated using population pharmacokinetic (PK) model. PK sparse sampling was performed. One sample was collected at anytime between 1 to 5 hours post-dose on Days 99 and 113 (Cohort 1, Cohort 2, Cohort 3) and two samples were collected, one at pre-dose and other at anytime between 1 to 5 hours post-dose on Days 99 and 113 (Cohort 4). Plasma concentrations of perampanel were measured and concentration data were summarized. Plasma concentrations of perampanel were quantified using a validated liquid chromatography mass spectrometry (LC MS/MS) analytical method.
Time Frame: Maintenance Period of the Core Phase- Days 99 and 113: 1-5 hours post-dose (Cohort 1, Cohort 2, Cohort 3); Days 99 and 113: Pre-dose, 1-5 hours post-dose (Cohort 4)
Population: The PK Analysis Set was the group of participants with at least 1 PK assessment of perampanel during the Maintenance Period (Core Phase) with a documented dosing history. Here, "overall number of participants analyzed" signifies participants who were evaluable for this Outcome Measure (OM).
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Groups:
- Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel (Non-EIAED): Participants of age range from >=1 to <=6 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to 12 mg/day (for participants who are not taking any EIAED). Dose titration was up to Week 12 for Non-EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose level 12 mg/day (for Non-EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase.
- Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel (Non-EIAED): Participants of age range from >6 to <=12 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to 12 mg/day (for participants who are not taking any EIAED). Dose titration was up to Week 12 for Non-EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose level 12 mg/day (for Non-EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase.
- Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel (Non-EIAED): Participants of age range from >12 to <24 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to 12 mg/day (for participants who are not taking any EIAED). Dose titration was up to Week 12 for Non-EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose level 12 mg/day (for Non-EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase.
- Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel (Non-EIAED): Participants of age range from >=24 to <48 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to 12 mg/day (for participants who are not taking any EIAED). Dose titration was up to Week 12 for Non-EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose level 12 mg/day (for Non-EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase.
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel (Non-EIAED) | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel (Non-EIAED) | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel (Non-EIAED) | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel (Non-EIAED)
Number analyzed (Participants) | 4 | 3 | 4 | 1
nanogram*hour per milliliter (ng*h/mL) | 3840 (2280) | 6110 (1490) | 6030 (1940) | 5810 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

23. Primary Outcome: Dose Normalized Maximum (Peak) Steady-state Concentration (Cmax,ss) of Perampanel During the Maintenance Period of the Core Phase for Non-EIAED Participants
Description: Dose normalized Cmax,ss was calculated as Cmax,ss/maintenance dose, where Cmax,ss is the maximum (peak) steady-state concentration calculated using population PK model. PK sparse sampling was performed. One sample was collected at anytime between 1 to 5 hours post-dose on Days 99 and 113 (Cohort 1, Cohort 2, Cohort 3) and two samples were collected, one at pre-dose and other at anytime between 1 to 5 hours post-dose on Days 99 and 113 (Cohort 4). Plasma concentrations of perampanel were measured and concentration data were summarized. Plasma concentrations of perampanel were quantified using a validated LC MS/MS analytical method.
Time Frame: as for outcome 22
Population: The PK Analysis Set was the group of participants with at least 1 PK assessment of perampanel during the Maintenance Period (Core Phase) with a documented dosing history. Here, "overall number of participants analyzed" signifies participants who were evaluable for this OM.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel (Non-EIAED) | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel (Non-EIAED) | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel (Non-EIAED) | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel (Non-EIAED)
Number analyzed (Participants) | 4 | 3 | 4 | 1
nanogram per milliliter (ng/mL) | 305 (73.1) | 388 (68.4) | 386 (103) | 341 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

24. Primary Outcome: Dose Normalized Average Steady-state Drug Concentration (Css,Av) of Perampanel During the Maintenance Period of the Core Phase for Non-EIAED Participants
Description: Dose normalized Css,Av was calculated as Css,Av/maintenance dose. Css,Av of perampanel was calculated as the ratio of area under the curve (AUC)/tau, (tau = 24 hours for perampanel) using population PK model. PK sparse sampling was performed. One sample was collected at anytime between 1 to 5 hours post-dose on Days 99 and 113 (Cohort 1, Cohort 2, Cohort 3) and two samples were collected, one at pre-dose and other at anytime between 1 to 5 hours post-dose on Days 99 and 113 (Cohort 4). Plasma concentrations of perampanel were measured and concentration data were summarized. Plasma concentrations of perampanel were quantified using a validated LC MS/MS analytical method.
Time Frame: as for outcome 22
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel (Non-EIAED) | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel (Non-EIAED) | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel (Non-EIAED) | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel (Non-EIAED)
Number analyzed (Participants) | 4 | 3 | 4 | 1
ng/mL | 160 (95) | 255 (62.2) | 251 (80.8) | 242 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

25. Primary Outcome: Dose Normalized Minimum Observed Steady State Plasma Concentration (Cmin,ss) of Perampanel During the Maintenance Period of the Core Phase for Non-EIAED Participants
Description: Dose normalized Cmin,ss was calculated as Cmin,ss/maintenance dose, where Cmin,ss is the minimum observed steady state plasma concentration calculated using population PK model. PK sparse sampling was performed. One sample was collected at anytime between 1 to 5 hours post-dose on Days 99 and 113 (Cohort 1, Cohort 2, Cohort 3) and two samples were collected, one at pre-dose and other at anytime between 1 to 5 hours post-dose on Days 99 and 113 (Cohort 4). Plasma concentrations of perampanel were measured and concentration data were summarized. Plasma concentrations of perampanel were quantified using a validated LC MS/MS analytical method.
Time Frame: as for outcome 22
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel (Non-EIAED) | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel (Non-EIAED) | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel (Non-EIAED) | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel (Non-EIAED)
Number analyzed (Participants) | 4 | 3 | 4 | 1
ng/mL | 114 (96.4) | 203 (58.2) | 199 (71) | 203 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

26. Primary Outcome: Dose Normalized AUCtau,ss of Perampanel During the Maintenance Period of the Core Phase for EIAED Participants
Description: Dose normalized AUCtau,ss was calculated as AUCtau,ss/maintenance dose, where AUCtau,ss is the area under the curve during a dosing interval (tau, 24 hours) at steady state calculated using population PK model. PK sparse sampling was performed. One sample was collected at anytime between 1 to 5 hours post-dose on Days 127 and 141 (Cohort 1, Cohort 2, Cohort 3) and two samples were collected, one at pre-dose and other at anytime between 1 to 5 hours post-dose on Days 127 and 141 (Cohort 4). Plasma concentrations of perampanel were measured and concentration data were summarized. Plasma concentrations of perampanel were quantified using a validated LC MS/MS analytical method.
Time Frame: Maintenance Period of the Core Phase- Days 127 and 141: 1-5 hours post-dose (Cohort 1, Cohort 2, Cohort 3); Days 127 and 141: Pre-dose, 1-5 hours post-dose (Cohort 4)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel (EIAED): Participants of age range from >=1 to <=6 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to 16 mg/day (for participants who are taking any EIAED). Dose titration was up to Week 16 for EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose level 16 mg/day (for EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase.
- Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel (EIAED): Participants of age range from >6 to <=12 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to 16 mg/day (for participants who are taking any EIAED). Dose titration was up to Week 16 for EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose level 16 mg/day (for EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase.
- Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel (EIAED): Participants of age range from >12 to <24 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to 16 mg/day (for participants who are taking any EIAED). Dose titration was up to Week 16 for EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose level 16 mg/day (for EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase.
- Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel (EIAED): Participants of age range from >=24 to <48 months received perampanel 0.5 mg, oral suspension, before bedtime during Week 0 and then dose up titrated to 16 mg/day (for participants who are taking any EIAED). Dose titration was up to Week 16 for EIAED participants to identify each participant's optimum dose during Core Phase. Participants then continued to take perampanel at optimal dose level 16 mg/day (for EIAED participants) as a maintenance dose for up to 4 weeks during Core Phase.
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel (EIAED) | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel (EIAED) | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel (EIAED) | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel (EIAED)
Number analyzed (Participants) | 0 | 2 | 3 | 1
ng*h/mL |  | 5220 (3600) | 3300 (1530) | 2510 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

27. Primary Outcome: Dose Normalized Cmax,ss of Perampanel During the Maintenance Period of the Core Phase for EIAED Participants
Description: Dose normalized Cmax,ss was calculated as Cmax,ss/maintenance dose, where Cmax,ss is the maximum (peak) steady-state concentration calculated using population PK model. PK sparse sampling was performed. One sample was collected at anytime between 1 to 5 hours post-dose on Days 127 and 141 (Cohort 1, Cohort 2, Cohort 3) and two samples were collected, one at pre-dose and other at anytime between 1 to 5 hours post-dose on Days 127 and 141 (Cohort 4). Plasma concentrations of perampanel were measured and concentration data were summarized. Plasma concentrations of perampanel were quantified using a validated LC MS/MS analytical method.
Time Frame: as for outcome 26
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel (EIAED) | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel (EIAED) | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel (EIAED) | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel (EIAED)
Number analyzed (Participants) | 0 | 2 | 3 | 1
ng/mL |  | 341 (151) | 276 (81.8) | 201 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

28. Primary Outcome: Dose Normalized Css,Av of Perampanel During the Maintenance Period of the Core Phase for EIAED Participants
Description: Dose normalized Css,Av was calculated as Css,Av/maintenance dose. Css,Av of perampanel was calculated as the ratio of area under the curve (AUC)/tau, (tau = 24 hours for perampanel) using population PK model. PK sparse sampling was performed. One sample was collected at anytime between 1 to 5 hours post-dose on Days 127 and 141 (Cohort 1, Cohort 2, Cohort 3) and two samples were collected, one at pre-dose and other at anytime between 1 to 5 hours post-dose on Days 127 and 141 (Cohort 4). Plasma concentrations of perampanel were measured and concentration data were summarized. Plasma concentrations of perampanel were quantified using a validated LC MS/MS analytical method.
Time Frame: as for outcome 26
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel (EIAED) | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel (EIAED) | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel (EIAED) | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel (EIAED)
Number analyzed (Participants) | 0 | 2 | 3 | 1
ng/mL |  | 217 (150) | 137 (63.8) | 105 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

29. Primary Outcome: Dose Normalized Cmin,ss of Perampanel During the Maintenance Period of the Core Phase for EIAED Participants
Description: Dose normalized Cmin,ss was calculated as Cmin,ss/maintenance dose, where Cmin,ss is the minimum observed steady state plasma concentration calculated using population PK model. PK sparse sampling was performed. One sample was collected at anytime between 1 to 5 hours post-dose on Days 127 and 141 (Cohort 1, Cohort 2, Cohort 3) and two samples were collected, one at pre-dose and other at anytime between 1 to 5 hours post-dose on Days 127 and 141 (Cohort 4). Plasma concentrations of perampanel were measured and concentration data were summarized. Plasma concentrations of perampanel were quantified using a validated LC MS/MS analytical method.
Time Frame: as for outcome 26
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel (EIAED) | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel (EIAED) | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel (EIAED) | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel (EIAED)
Number analyzed (Participants) | 0 | 2 | 3 | 1
ng/mL |  | 172 (145) | 90.5 (53.4) | 69.2 (NA) — Standard Deviation could not be calculated as only one participant was available for analysis.

ADVERSE EVENTS:
Time Frame: Core Phase: From the first dose of study drug up to 4 weeks of follow up after the last dose in Core Phase (up to Week 24); Extension Phase: From end of Core Phase treatment up to 4 weeks of follow up after the last dose in Extension Phase (up to Week 56)
Description: The SAS was the group of participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment.
Arm/Group | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5 | 0/9 | 0/3 | 0/4 | 0/5 | 0/8 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/5 | 2/9 | 1/3 | 3/4 | 1/5 | 3/8 | 0/1
Other Adverse Events (participants affected / at risk) | 2/4 | 5/5 | 9/9 | 2/3 | 2/4 | 5/5 | 8/8 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel (N=4) | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel (N=5) | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel (N=9) | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel (N=3) | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel (N=4) | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel (N=5) | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel (N=8) | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel (N=1)
Bullous impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 1 (2) | 2 (5) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenovirus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterovirus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure To Thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel (N=4) | Core Phase, Cohort 2, Age >6 to <=12 Months: Perampanel (N=5) | Core Phase, Cohort 3, Age >12 to <24 Months: Perampanel (N=9) | Core Phase, Cohort 4, Age >=24 to <48 Months: Perampanel (N=3) | Extension Phase, Cohort 1, Age >=1 to <=6 Months: Perampanel (N=4) | Extension Phase, Cohort 2, Age >6 to <=12 Months: Perampanel (N=5) | Extension Phase, Cohort 3, Age >12 to <24 Months: Perampanel (N=8) | Extension Phase, Cohort 4, Age >=24 to <48 Months: Perampanel (N=1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (4) | 3 (4) | 1 (2) | 0 (0) | 2 (4) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (8) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 0 (0)
Lip Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 5 (9) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (2)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food Allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia Aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotavirus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oxygen Saturation Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Failure To Thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Status Epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Device Dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenoidal Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-09): https://cdn.clinicaltrials.gov/large-docs/14/NCT02914314/Prot_002.pdf
  • Statistical Analysis Plan (2023-02-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT02914314/SAP_003.pdf